CLINICAL TRIAL: NCT03141788
Title: Evaluation of 3M Clear Aligner for Correction of Class I, II and III Malocclusion Study
Brief Title: Evaluation of Clear Aligner Trays to Straighten Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum Orthodontics Corporation (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US-05-013821/11-050005
Record Dates: First submitted 2017-04-27; First posted 2017-05-05 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Malocclusion
Keywords: Aligners
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 3M Clear Aligner (Other): Clear Aligner for Orthodontic Treatment
  Interventions: Device: Clear Aligner

INTERVENTIONS:
Device: Clear Aligner — Clear Aligner used to straighten teeth to desired outcome
  Other Names: 3M Clear Aligner

SUMMARY:
The objective of this study is to evaluate the efficacy of Clear Aligners to correct tooth malocclusions with the use of attachments and/or buttons, as determined by the amount of teeth movement and overall achievement goals of the treatment plan.

DETAILED DESCRIPTION:
This is a prospective, multi-center study with a maximum duration of 24 months or longer depending on refinements, to assess the safety and efficacy of 3M Clear Aligners, with the use of attachments to correct teeth malocclusions.

The subject population for this study will be male and female subjects ≥ 14 years of age. Subjects who meet the inclusion and exclusion criteria will be asked to participate in the study. Up to a total of 180 subjects may be enrolled at up to 12 different clinical research sites, (up to 15 subjects per site).

The subjects will undergo a target of up to 24 months (or longer depending on refinements) of treatment to align the teeth to the planned target. Subjects will wear the Clear Aligners for at least 22 hours per day, with the exception of consumption of meals and beverages, with the exception of water, which can be consumed while wearing the aligners. During each 6-week period between follow up visits, subjects will wear each set of Clear Aligners for 2 weeks, in the order indicated per the Orthodontists treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 14 years of age.
2. Subject is willing and able to give informed consent.
3. Subject is willing to be digitally scanned at each 6-week visit, including after application of attachments.
4. Subject has a need for single or double arch orthodontic treatment with a target duration of 18 months or less.
5. Subject has good oral hygiene defined by the orthodontist.
6. Subject has only permanent dentition.

Exclusion Criteria:

1. Subject has skeletal discrepancies requiring surgery
2. Subject is undergoing active dental work
3. Subject has severe open bite > 2 mm
4. Subject has severe overjet > 4 mm
5. Subject has deep bite > 3 mm
6. Subject has over crowding per arch > 4 mm
7. Subject has dental prostheses/implants that will interfere with projected teeth movement
8. Subject is taking systemic steroid medication
9. Subject is taking Biphosphonates or any other medication for treatment of osteoporosis

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail E Maxey, BA, CCRA, Study Director — 3M Company
Locations (9):
- United States (9):
  - Benson Orthodontics, Denver, Colorado
  - Depew Orthodontics, Kennesaw, Georgia
  - Orthodontics Associates, Catonsville, Maryland
  - Henseler Orthodontics, Woodbury, Minnesota
  - Horton Orthodontics, Woodbury, Minnesota
  - Mellion Orthodontics, Fairlawn, Ohio
  - Wolf/Chhibber Orthodontics, Norwalk, Ohio
  - Simply Smiles Orthodontics, McKinney, Texas
  - Riolo Orthodontics, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screen failures because they did not meet Inclusion/Exclusion criteria
Groups:
- 3M Clear Aligner: 3M Clear Aligner for Orthodontic Treatment
Period: Overall Study
Arm/Group | 3M Clear Aligner
Started | 52
Completed | 44
Not Completed | 8
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- 3M Clear Aligner: Clear Aligner Treatment
  Clear Aligner: Clear Aligner used to straighten teeth to desired outcome
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 46
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 52
Class type of malocclusion [Count of Participants; unit: Participants] — Class I Malocclusion - the bite is normal but the upper teeth slightly overlap the lower teeth
  Class II Malocclusion - the upper jaw and teeth severely overlap the bottom jaw and teeth (overbite)
  Class III Malocclusion - the lower jaw is advanced forward or the upper jaw is held back (underbite)
  Participants
    Class I Malocclusion | 39
    Class II Malocclusion | 12
    Class III Malocclusion | 1
Previous orthodontic treatments [Count of Participants; unit: Participants]
  Yes | 32
  No | 20

OUTCOME MEASURES:

1. Primary Outcome: Successful Correction of Malocclusion
Description: Achievement of target setup per treatment plan as determined by Orthodontist.
Time Frame: The expected duration of subject participation was to be 6 to 24 months. Due to additional time needed for orthodontic refinements, the actual longest duration was approximately 28 months.
Measure: Count of Participants; unit: Participants
Groups:
- 3M Clear Aligner: Clear Aligner Orthodontic Treatment for malocclusion
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Participants
  Reached Target Set Up | 32
  Did Not Reach Target Set Up | 20

2. Secondary Outcome: Individual Tooth Movement
Description: Achievement of individual tooth movement measured per treatment plan and digital scan
Time Frame: as for outcome 1
Population: Not obtained due to technical difficulties including warped and insufficient dental scans
Groups:
- 3M Clear Aligner: Clear Aligner Orthodontic Treatment
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 0

3. Secondary Outcome: Treatment Time for Tooth Movement
Description: Achievement of individual tooth movement measured per treatment plan
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
days | 443 [14 to 853]

4. Secondary Outcome: Effective Use of Attachments
Description: Effective use of attachment by tracking attachment bond failures by visual assessment
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Attachment Bond Failure
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Percentage of Attachment Bond Failure | 5.4 (14.58)

5. Secondary Outcome: Orthodontist Satisfaction
Description: Orthodontist satisfaction with treatment outcome
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Participants
  Very Satisfied | 5
  Satisfied | 33
  Neutral | 7
  Dissatisfied | 2
  Not Applicable | 5

6. Secondary Outcome: Software Satisfaction
Description: Orthodontist satisfaction with treatment management software -Ease of use in ordering products
Time Frame: as for outcome 1
Population: The ordering software was updated during treatment and therefore not analyzed.
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 0

7. Secondary Outcome: Aligner Comfort
Description: Aligner comfortable to wear
Time Frame: as for outcome 1
Measure: Count of Units; unit: study visits
Units Other Than Participants: study visits
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Number analyzed (study visits) | 479
study visits
  Extremely Comfortable | 24
  Comfortable | 390
  Tolerable | 41
  Somewhat Uncomfortable | 22
  Not at all Comfortable | 2

8. Secondary Outcome: Appearance Satisfaction
Description: Subject satisfaction with appearance during treatment
Time Frame: as for outcome 1
Measure: Count of Units; unit: study visits
Units Other Than Participants: study visits
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Number analyzed (study visits) | 479
study visits
  Satisfied | 470
  Not Satisfied | 9

9. Secondary Outcome: Aligner Ease of Cleaning
Description: Subject satisfaction with ease of cleaning during treatment
Time Frame: as for outcome 1
Measure: Count of Units; unit: study visits
Units Other Than Participants: study visits
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Number analyzed (study visits) | 479
study visits
  Easy to Keep Clean | 436
  Not Easy to Keep Clean | 43

10. Secondary Outcome: Ease of Insertion
Description: Subject satisfaction with treatment; specifically aligners easy to insert
Time Frame: as for outcome 1
Measure: Count of Units; unit: study visits
Units Other Than Participants: study visits
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Number analyzed (study visits) | 479
study visits
  Easy | 364
  Somewhat Easy | 97
  Somewhat Difficult | 15
  Difficult | 3

11. Secondary Outcome: Mid Course Corrections/Refinements Needed
Description: Number of mid course refinements or corrections
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Participants
  No Corrections/Refinements | 21
  1 Corrections/Refinements | 19
  2 Corrections/Refinements | 8
  3 Corrections/Refinements | 4

12. Secondary Outcome: Ease of Aligner Removal
Description: Subject satisfaction with treatment; specifically with aligner removal
Time Frame: as for outcome 1
Measure: Count of Units; unit: study visit
Units Other Than Participants: study visit
Arm/Group | 3M Clear Aligner
Number analyzed (Participants) | 52
Number analyzed (study visit) | 479
study visit
  Easy | 308
  Somewhat Easy | 136
  Somewhat Difficult | 32
  Difficult | 3

ADVERSE EVENTS:
Time Frame: Up to 28 months
Arm/Group | 3M Clear Aligner
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3M Clear Aligner (N=52)
Bleeding Gums (Gastrointestinal disorders) | 1 (1) — Bleeding Gums
Filling Fell Off Tooth (Product Issues) | 1 (2) — Filling Fell Out of Tooth

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03141788/Prot_SAP_000.pdf